CLINICAL TRIAL: NCT02140398
Title: Endometrial Scratching at Time of Laproscopic Ovarian Drilling in Women With Anovulatory Infertility Due to Polycystic Ovarian Syndrome (PCOS): Randomized Controlled Trial.
Brief Title: Endometrial Scratching During Laproscopic Ovarian Drilling in Subfertile PCOS Women
Acronym: ESLOD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Gibreel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 92013
Record Dates: First submitted 2014-04-25; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Infertility; Polycystic Ovarian Syndrome
Keywords: infertility; PCOS; scratching; endometrial receptivity
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Currettage (Experimental): Endometrial Currettage (endometrial scrapping) will be performed at the time of laparoscopic ovarian drilling
  Interventions: Procedure: Endometrial Currettage
- Nothing (No Intervention): No endometrial curettage at time of Laparoscopic ovarian drilling

INTERVENTIONS:
Procedure: Endometrial Currettage — Only Laparoscopic ovarian drilling without endometrial currettage will be performed
  Other Names: Endometrial injury; endometrial scratching; Endometrial scraping
  Arms: Currettage

SUMMARY:
Laparoscopic Ovarian Drilling is a valid procedure for infertile anovulatory women with polycystic ovarian syndrome who failed to get pregnant or to ovulate with ovulation induction medications as clomiphene citrate or exogenous gonadotropins. The reasearchers supposed that endometrial curettage at time of laparoscopic ovarian drilling may boost fertility in these women.

DETAILED DESCRIPTION:
Current literature suggests that endometrial biopsy may improve pregnancy rates in infertile women hence the investigators will examine whether this hypothesis will apply to infertile PCOS women undergoing laparoscopic ovarian drilling to overcome ovulatory disfunction or not.

ELIGIBILITY:
Inclusion Criteria:

1. subfertile women with anovulatory infertility due to polycystic ovarian syndrome (PCOS).
2. Women who failed to get pregnant after at least 6 months of ovulation induction cycles with clomiphene citrate or exogenous gonadotropins
3. Patent Fallopian tubes as confirmed by hysterosalpingography
4. Fertile semen parameters of the partneraccording to criteria of World Health Organization (WHO 2010).

Exclusion Criteria:

1. women with BMI >30,
2. age < 18 years or > 39 years,
3. women with ovarian cysts identified by transvaginal ultrasound
4. male factor infertility
5. Tubal factor infertility as suggested by hystrosalpingogram (HSG)
6. Women with congenital malformations in the uterus as bicornuate or septate uterus as suggested by HSG.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
live birth rate per woman randomized | 15 months

SECONDARY OUTCOMES:
pregnancy rate per woman randomised | 6 months

OTHER OUTCOMES:
miscarriage rate time to pregnancy interval | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gibreel, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Teaching Hospital, Al Mansurah, Egypt